CLINICAL TRIAL: NCT01093352
Title: The Efficacy of Surgical Exposure With Alveolar-decortication vs. Conventional Surgical Exposure to Reduce Treatment Time for Orthodontic Alignment of Palatally Impacted Canines
Brief Title: Effect of Alveolar-decortication on Velocity of Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, Mary Alice Bussell, SpR in orthodontics, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09/H1207/108
Record Dates: First submitted 2010-03-18; First posted 2010-03-25 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Palatally Impacted Canines
Keywords: Alveolar-decortication; Corticotomy assisted orthodontics; Palatally impacted canine; Surgical exposure of canines; Velocity of tooth movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (No Intervention): Standard expose and bond.
- Alveolar-decortication (Experimental): Following surgical exposure of the impacted canine, additional perforations will be made in the surrounding cortical bone prior to wound closure.
  Interventions: Procedure: Alveolar-decortication.

INTERVENTIONS:
Procedure: Alveolar-decortication. — Following surgical exposure of the impacted tooth, the surgeon will prepare small holes (perforations) and/or grooves in the cortical bone surrounding the exposed tooth as well as in the buccal bone.
  Other Names: Alveolar-decortication; Corticotomy assisted orthodontics
  Arms: Alveolar-decortication

SUMMARY:
The purpose of this pilot clinical trial is to evaluate whether alveolar-decortication has the potential to reduce orthodontic treatment time following surgical exposure of palatally impacted canines.

DETAILED DESCRIPTION:
Purpose:

Upper permanent canines frequently become impacted (2%), which prevents their normal eruption (Brin et al, 1986. Ericson and Kurol, 1986). The upper canine may become impacted palatally (61%) or buccally (4.5%) (Stivaros and Mandall, 2000).

One of the treatment options for impacted canines is to surgically expose the canine tooth and to align it using orthodontic appliances. A bracket is attached to the tooth at the time of surgery. The tooth is then aligned using orthodontic forces.

Alveolar-decortication is also referred to as corticotomy-assisted orthodontics (Fischer, 2007). The technique involves exposure of alveolar bone and partial decortication of the cortical plates followed by primary flap closure.

It is believed that this alternative surgical technique reduces the time taken to orthodontically align teeth; previous case reports and preliminary studies report reductions by 28% to 80% in treatment time (Fischer, 2007. Wilcko et al, 2001).

No rigorous clinical trials have been conducted to evaluate the efficacy of alveolar-decortication to reduce orthodontic treatment times. We plan to evaluate this technique in patients with palatally impacted canines because a surgical procedure is necessary anyway to expose the tooth and the additional surgical trauma is minimal.

Aims and objectives:

This study aims to investigate the effect of alveolar-decortication in addition to surgical exposure, on the time taken to align palatally impacted canines. The alternative surgical technique will be compared to the conventional surgical exposure, by recording the time taken to subsequently align the tooth.

The objective is to determine whether the use of alveolar-decortication whilst exposing an impacted tooth, will lead to a reduction in the time required to align the tooth, and therefore a reduction in the overall treatment time.

Recruitment and consent:

30 orthodontic patients (n=15 per group), who are awaiting exposure and bonding of a palatally impacted canine tooth, will be selected from the waiting list at Birmingham Dental Hospital. Potential participants will be invited to take part in the study; they will be given verbal and written information. If they are happy to take part, written consent will be obtained. All patients recruited will be competent and capable of making the decision. For patients under 16 years of age, parental/legal guardian consent will be obtained. The patients will be able to withdraw from the study at any time, should they not wish to continue participating.

Methods:

Participants will be randomly allocated to either the control or test group, at the time of surgery.

Randomisation will use the method of randomly permuted blocks with variable block size. Enrolled participants will be assigned a study number at the time of surgery. The envelope with group assignment will be opened after completion of the surgical exposure (prior to wound closure). For subjects randomised to the test group, alveolar-decortication will then be carried out prior to wound closure. While the surgeon cannot be blinded for obvious reasons, group assignment will not be disclosed to the patient and will not be disclosed to the orthodontist.

At the time of surgery, 3 intra-oral photographs will be taken of the upper arch, including the exposed tooth.

Following surgery, the orthodontic treatment will be carried out in the normal way. At routine appointments, 3 intra-oral photographs will be taken of the upper arch, including the canine tooth. These photographs will be inserted into a computer programme, and a stereo-imaging technique will be used to construct a 3-D image, which will allow the velocity of tooth movement to be calculated.

Impressions will be taken of the upper arch during treatment, the resultant study models can also be used to calculate velocity of tooth movement. The distance between the tip of the canine tooth, to the line of the arch will be measured with callipers, at the time of surgery and also during routine orthodontic appointments.

Inclusion criteria:

Patients at Birmingham Dental Hospital. Patients with a palatally impacted canine, awaiting surgical exposure. Patients with bilateral impacted canines may be included, in these cases both canines will be treated using the same surgical technique determined by allocation into either the test or control group.

Informed consent gained.

Exclusion criteria:

History of periodontal disease. Radiographical evidence of pathology associated with the impacted canine. Patients already participating in a research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Birmingham Dental Hospital.
* Patients with a palatally impacted canine, awaiting surgical exposure.
* Patients with bilateral impacted canines may be included; in these cases both canines will be treated using the same surgical technique determined by allocation into either the test or control group.
* Informed consent gained.

Exclusion Criteria:

* History of periodontal disease.
* Radiographical evidence of pathology associated with the impacted canine.
* Patients already participating in a research study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02-23 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Velocity of tooth movement | 6-8 weeks
  The velocity of movement of the canine tooth will be recorded, from the start (buried) position until it is in the line of the arch. Measurements will be taken at each orthodontic appointment, usually 6-8 weeks apart throughtout treatment.
  Distance will be measured with the use of linear measurements, impressions and clinical photographs.

SECONDARY OUTCOMES:
Time for alignment | approx. 2 years.
  This will record the overall time for canine alignment, from its initial position to its final position when active orthodontic appliances are removed.
Total orthodontic treatment time | approx. 2.5 years.
  This will record the overall time, from placement to removal of active orthodontic appliances.
Duration of surgery | 1 day
  The duration of the surgical procedure in minutes, the time inbetween raising and closing the flap of gum tissue will be recorded.
Adverse effects of surgery | approx. 2.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, DMD, MD, MPH, Principal Investigator — School of Dentistry, University of Birmingham.
Locations (1):
- School of Dentistry, University of Birmingham, Birmingham, United Kingdom